CLINICAL TRIAL: NCT04749056
Title: Evaluation of an Electronic Psycho-oncological Adaptive Screening Program to Assess Psychological Burden and Need for Psycho-social Support Among Cancer Patients
Brief Title: Electronic Psycho-oncological Adaptive Screening Program
Acronym: EPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hamburg-Eppendorf (Other)
Collaborators: Federal Ministry of Health, Germany (Other Government); University of Leipzig (Other)
Responsible Party: Principal Investigator, Anja Mehnert, Prof. Dr. Anja Mehnert-Theuerkauf, University of Leipzig
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EPAS_Intervention
Record Dates: First submitted 2021-01-25; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Non-randomized controlled evaluation study (cluster crossover design) to test a screening program to assess psychological burden and supportive care needs among cancer patients.
  Patients undergoing the screening (intervention group) will be compared to patients without the screeninig (control group).
  The study has three measurement points: T0 (before the intervention), T1 (3 months after the intervention) and T2 (6 months after the intervention). Care relevant outcomes which are not yet relevant at T0 (information level, use of psychosocial services, treatment satisfaction) will be assessed at T1 and T2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPAS screening (intervention) (Experimental): Patients undergo EPAS (electronic psycho-oncological adaptive screening), a tablet-based screening application consisting of three adaptive tests and one supportive care checklist. EPAS provides immediate feedback via a printed results page, which presents and interprets the level of distress and contains individualized recommendations for psychosocial services.
  The results pages are printed by research assistants immediately after the screening on a mobile printer and given to the participants together with a brochure containing information about all psychosocial services available at the health care institution.
  The treating physicians also receive a slightly modified results page, but are not expected to discuss these with the patient unless they are highly distressed.
  Before and during the screening, patients are explained how to use the program by the research assistance and supported if needed.
  The whole screening process takes about 30 minutes.
  Interventions: Behavioral: EPAS (electronic psycho-oncological adapative screening program)
- Care as usual (control) (No Intervention): Patients complete the assessment paper pencil. The same instruments as in the intervention condition are used except for the 3 adaptive tests (i.e., the supportive care checklist and the outcomes).
  Neither patients nor physicians receive any feedback of the results. Psychosocial services are recommended by the physicians on their own discretion only, and patients are not handed out the information brochure.

INTERVENTIONS:
Behavioral: EPAS (electronic psycho-oncological adapative screening program) — Adaptive tests assess depression, anxiety and distress. Only items with highest information value are selected. Furthermore, patients fill in a checklist to report supportive care needs.
  The results page contains (i) the extent of distress and additional information to interpret these levels, (ii) a summary of the reported supportive care needs and (iii) individualized recommendations for the use of psychosocial services at the institution based on the care needs.
  The supportive care needs are transformed into concrete recommendations to use the adequate psychosocial service at the institution. Highly distressed patients are recommended to use psycho-oncological service irrespective of whether they have reported such a need in the check list. Physicians of highly distressed patients are recommended on their results page to talk with the patient about his/her psychosocial condition and further issues within such an appointment are suggested.
  Arms: EPAS screening (intervention)

SUMMARY:
Background: Psychological burden in cancer patients may worsen quality of life and even medical outcomes such as mortality. Nevertheless, many distressed patients are not recognized by the treating clinicians and left untreated even though effective psychosocial interventions exist. Existing screenings programs have multiple limitations such as the necessity of time consuming training and involvement of clincial staff, conventional screening instruments with limited diagnostic accuracy and the focusing on objective measures of distress, thereby neglecting subjective supportive care needs.

Aims: To address some of the limitations outlined above, we developed an electronic psycho-oncological adaptive screening program (EPAS) which separately assesses distress and psychosocial care needs and provides immediate patient feedback with individualized recommendations about psychosocial care services.

Design: Patients of the intervention are compared to a control condition. All participants are assessed at three measurement points (baseline, and at 3-months and 6-months follow-up).

Outcomes: Outcomes assess aspects related to psychosocial care services, well-being and satisfaction.

Recruitment: Patients are recruited within suitable health care facilities within the University Cancer Center Hamburg (UCCH) and other facilities in the competence network of the UCCH. Patients are checked for eligibility via review of the medical chart and consecutively recruited by research assistants.

Duration of the study: From start of recruitment, 2 years are planned until data analysis. 1 year is planned for recruitment.

Analyses: We conduct group comparisons in the study outcomes, both unconditional and condcitional (controlled for care relevant co-variates).

DETAILED DESCRIPTION:
Background: Psychological burden in cancer patients may worsen quality of life and even medical outcomes such as mortality. Nevertheless, many distressed patients are not recognized by the treating clinicians and left untreated even though effective psychosocial interventions exist. Existing screenings in turn have multiple limitations: To be effective in reducing distress, screening results need to be adequately interpreted and transformed into individualized support plans. Most of current screening programs expect the clinical staff to undertake this task, which in turn requires extensive and repeated training. Another critical issue is the assessment: To limit the completion time to a minimum, conventional screening instruments contain as few items as possible, which in turn limits their diagnostic accuracy. Finally, most screening programs assume that there is a clear link between reported levels of distress and the individual need for psychosocial care. Accordingly, many current screenings derive the need for psychosocial care exclusively from the level of distress reported by the patients. However, self-reported distress and self-reported supportive care need are not closely related.

Aims of the study: To address some of the limitations outlined above, we developed an electronic psycho-oncological adaptive screening program (EPAS) which separately assesses distress and psychosocial care needs and provides immediate patient feedback with individualized recommendations about psychosocial care services.

Design: Patients of the intervention are compared to a control condition. All participants are assessed at three measurement points (baseline, and at 3-months and 6-months follow-up).

Outcomes: Outcomes assess aspects related to psychosocial care services, well-being and satisfaction.

Sample size: Our study aims to separately test for group differences (screening vs. no screening) at t1 and t2. To detect an expected small to medium group difference in level of information (effect size = 0.3) with a power of 80 %, sample sizes of 176 patients in each group were needed. Given an expected drop-out rate of 30 % from t0 to t2, we initially planned to recruit n = 251 per group (ntotal = 502).

Recruitment: Patients are recruited within suitable health care facilities within the University Cancer Center Hamburg (UCCH) and facilities in the competence network of the UCCH. Patients are checked for eligibility via review of the medical chart and consecutively recruited by research assistants.

Sample: We applied a cross-over design: That is, all clusters received each intervention so that a largely equal number of patients received each intervention in each cluster. Between the changes of the conditions, recruitment was suspended for a certain amount of time to avoid any overlap of patients in the two conditions.

Duration of the study: From start of recruitment, 2 years are planned until data analysis. 1 year is planned for recruitment.

Analyses: We conduct group comparisons in the study outcomes separately for t1 and t2. Robustness of the analyses is checked by calculating both unconditional and conditional (controlled for care relevant co-variates) models. In detail, we apply linear and logistic regression analyses for continous and binary outcomes, respectively.

Detailed description of the intervention:

General principle and procedure: The patients in the intervention arm undergo EPAS (electronic psycho-oncological adaptive screening), a tablet-based screening application consisting of three adaptive tests and one supportive care checklist. EPAS provides immediate feedback via a printed results page, which presents and interprets the level of distress and contains individualized recommendations for psychosocial services. The results pages are printed by research assistants immediately after the screening on a mobile printer and given to the participants together with a brochure containing information about all psychosocial services available at the UCCH. The treating physicians also receive a slightly modified results page, but are not expected to discuss these with the patient unless they are highly distressed (see algorithm section). Before and during the screening, patients are explained how to use the program by the research assistance and supported if needed. The whole screening process including the conventional tests that are also assessed by the control group takes about 30 minutes.

Measures within EPAS: Three adaptive tests with varying response options are applied to assess depression (D-CAT, 64 items), anxiety (A-CAT, 50 items) and distress/stress reaction (S-CAT, 38/31 items). From the item pools, only items with highest information value are selected according to both item characteristics and individual response pattern. The presentation of items ends if (i) the standard error was ≤ 0.32 or (ii) a maximum of 10 items is reached. Furthermore, patients fill in an internally developed checklist to report supportive care needs.

Structure and content of the results page: The results page contains (i) the extent of distress and additional information to interpret these levels, (ii) a summary of the reported supportive care needs and (iii) individualized recommendations for the use of psychosocial services at the UCCH based on the care needs. As additional information to interpret the levels of distress, categories derived from a psychosomatic population are provided for D-CAT and A-CAT (low/medium/high). No such categories exist for the S-CAT, and thus the mean among a population with burnout-syndrome is provided as a reference value. The patient and physician versions slightly differ: Whereas patients are explicitly referred to the information brochure they receive during the screening, the distress-categories in the physician version are illustrated with colors (low = green; medium = yellow; high = red) and contain specific information in case of highly distressed patients (see algorithm section).

Algorithm for the results page: The supportive care needs reported in the respective list are transformed into concrete recommendations to use the adequate psychosocial service at the UCCH (e.g., a reported need for support to return to work results in a recommendation to use the social service). Highly distressed patients, i.e., those falling in the category "high" in the A-CAT or D-CAT, are recommended to use psycho-oncological service irrespective of whether they have previously reported such a need in the check list. Physicians of highly distressed patients are recommended on their results page to talk with the patient about his/her psychosocial condition and further issues within such an appointment are suggested (e.g., check for medical reasons for distress, encourage patients to use psycho-oncological service).

ELIGIBILITY:
Inclusion Criteria:

* minimum age of 18 years
* diagnosed with any malignancy according to ICD-10 (first diagnosis or relapse)

Exclusion Criteria:

* Patients with any impairments interfering with the ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Information level about psychosocial services at 3 months-follow-up | The outcome is assessed at T1 (3-months follow-up).
  On 10 items, patients rate their level of information for each of the 10 available psychosocial services on a scale from 0 to 4, with higher values indicating a higher level of information. Items are evaluated as single scales.
Information level about psychosocial services at 6 months-follow-up | The outcome is assessed at T2 (six months follow-up).
  On 10 items, patients rate their level of information for each of the 10 available psychosocial services on a scale from 0 to 4, with higher values indicating a higher level of information. Items are evaluated as single scales.
Use of the psychosocial services at 3-months follow-up | The outcome is assessed at T1 (3-months follow-up).
  On an internally developed questionnaire, patients rate on 10 binary items (yes/no) whether they have used each of the 10 psychosocial services available at the study center. The items are analysed as single scales.
Use of the psychosocial services at 6-months follow-up | The outcome is assessed at T2 (six months follow-up).
  On an internally developed questionnaire, patients rate on 10 binary items (yes/no) whether they have used each of the 10 psychosocial services available at the study center. The items are analysed as single scales.
Evaluation of access to psychosocial services | The outcome is assessed at T1 (3-months follow-up).
  On 4 nominal items (yes/no/do not know), we assess whether any i) communication with the physicians about supportive/complementary care needs, ii) recommendations by the physicians for psychosocial services, iii) concrete offers by the physicians to use a psychosocial service or iv) request by the physicians for a consultation service have taken place.
Depressive symptomatology at 3-months follow-up | The outcome is assessed at T1 (3-months follow-up).
  PHQ-9: On 9 items, patients rate the frequency of depressive symptoms on a scale from 0 to 3, with higher scores indicating a higher symptomatology (range of sum score: 0 - 27).
Depressive symptomatology at 6-months follow-up | The outcome is assessed at T2 (six months follow-up).
  PHQ-9: On 9 items, patients rate the frequency of depressive symptoms on a scale from 0 to 3, with higher scores indicating a higher symptomatology (range of sum score: 0 - 27).
Anxious symptomatology at 3-months follow-up | The outcome is assessed at T1 (3-months follow-up).
  GAD-7: On 7 items, patients rate the frequency of anxious symptoms on a scale from 0 to 3, with higher values indicating higher level of anxiety (range of sum score: 0 - 21).
Anxious symptomatology at 6-months follow-up | The outcome is assessed at T2 (6-months follow-up).
  GAD-7: On 7 items, patients rate the frequency of anxious symptoms on a scale from 0 to 3, with higher values indicating higher level of anxiety (range of sum score: 0 - 21).
Health-related quality of life at 3-months follow-up | The outcome is assessed at T1 (3-months follow-up).
  SF-8: On 8 items, patients rate their impairments of health-related quality of life across different areas on items ranging from 0 to 5/6. Items are later transformed on a scale from 0 to 100, with higher values indicating a higher level of quality of life.
Health-related quality of life at 6-months follow-up | The outcome is assessed at T2 (6-months follow-up).
  SF-8: On 8 items, patients rate their impairments of health-related quality of life across different areas on items ranging from 0 to 5/6. Items are later transformed on a scale from 0 to 100, with higher values indicating a higher level of quality of life.
Treatment satisfaction at 3-months follow-up | The outcome is assessed at T1 (3-months follow-up).
  On 32 items, patients rate their satisfaction with medical and psychosocial cancer care on a scale ranging from 1 to 5/6, with higher scores indicating higher level of satisfaction. The questionnaire is analysed by sum scores across specific subscales (Competence, Information, Access, Support, Overall medical treatment, Overall psychosocial treatment).
Treatment satisfaction at 6-months follow-up | The outcome is assessed at T2 (6-months follow-up).
  On 32 items, patients rate their satisfaction with medical and psychosocial cancer care on a scale ranging from 1 to 5/6, with higher scores indicating higher level of satisfaction. The questionnaire is analysed by sum scores across specific subscales (Competence, Information, Access, Support, Overall medical treatment, Overall psychosocial treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Anja Mehnert-Theuerkauf, Prof., Principal Investigator — University of Leipzig

REFERENCES:
- [Derived] Springer F, Sautier L, Schilling G, Koch-Gromus U, Bokemeyer C, Friedrich M, Mehnert-Theuerkauf A, Esser P. Effect of depression, anxiety, and distress screeners on the need, intention, and utilization of psychosocial support services among cancer patients. Support Care Cancer. 2023 Jan 16;31(2):117. doi: 10.1007/s00520-023-07580-2. PMID 36645499
- [Derived] Esser P, Sautier L, Sarkar S, Schilling G, Bokemeyer C, Koch U, Rose M, Friedrich M, Nolte S, Walter O, Mehnert-Theuerkauf A. Evaluation of an electronic psycho-oncological adaptive screening program (EPAS) with immediate patient feedback: findings from a German cluster intervention study. J Cancer Surviv. 2022 Dec;16(6):1401-1413. doi: 10.1007/s11764-021-01121-8. Epub 2021 Nov 4. PMID 34735695